CLINICAL TRIAL: NCT03995030
Title: Massively Parallel Sequencing to Identify Microbiological Organisms in Bronchoalveolar Lavage Fluid in Children, Adolescents and Young Adults Post Hematopoietic Stem Cell Transplant
Brief Title: Massively Parallel Sequencing to Identify Microbiological Organisms in Bronchoalveolar Lavage Fluid
Status: Completed | Type: Observational
Sponsor: New York Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: NYMC 181
Record Dates: First submitted 2019-06-06; First posted 2019-06-21 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Pulmonary Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extra BAL fluids will be sent to for massively parallel sequencing research tests at New York Medical College Genomics Core Facility.
  The research portion will be further divided for isolation of viral, bacterial, and fungal nucleic acid isolation. A control sample of fluid used for the BAL will be prepared in parallel. Bacterial/fungal DNA and viral DNA and RNA will be isolated. Whole genome sequencing libraries will be generated and sequenced in batches on the Illumina MiSeq.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: massively paralleled sequencing — Whole genome sequencing libraries will be generated and sequenced in batches on the Illumina MiSeq. FASTQ files will be demultiplexed and then aligned to microbial genomes using Phylosift.

SUMMARY:
Patients who are post hematopoietic stem cell transplantation who require a bronchoalveolar lavage (BAL) for standard clinical car will have extra fluid collected and sent for massively parallel sequencing to see if it is as sensitive for detecting a microbial pulmonary infection compared to standard cultures.

DETAILED DESCRIPTION:
5.1 Subjects will undergo bronchoscopy and BAL based on clinical indications. Techniques and equipment will be per current clinical practice at Westchester Medical Center (WMC). The bronchoscope is usually introduced either via an artificial airway (endotracheal tube or laryngeal mask airway). The lavage is performed with sterile normal saline. The site of performing the lavage is selected based on radiologic or clinical data and on the appearance of the airways during the bronchoscopy. The typical volume of the lavage is 3 aliquots of 1 ml/kg each, with a max of 20 ml per aliquot.

5.2 When 10 ml or more of BAL fluid is received by the WMC laboratory, the BAL fluid will be divided by the WMC laboratory for all physician ordered clinical laboratory tests and for massively parallel sequencing research tests. This will ensure that sufficient BAL material is available for all clinical tests.

5.3 The BAL fluid for research will be held by the WMC laboratory and picked up by research personnel for processing at New York Medical College Genomics Core Facility.

5.4 The research portion will be further divided for isolation of viral, bacterial, and fungal nucleic acid isolation. A control sample of fluid used for the BAL will be prepared in parallel. Bacterial/fungal DNA and viral DNA and RNA will be isolated. Whole genome sequencing libraries will be generated and sequenced in batches on the Illumina MiSeq.

FASTQ files will be demultiplexed and then aligned to microbial genomes using Phylosift.11 DNA sequences present in both the patient and control samples will be discarded as contaminant. The preponderant organism(s) identified will be matched to the results of the culture based techniques used to verify the culture independent results.

ELIGIBILITY:
Inclusion criteria

* Patient age < 30 years
* Recipient of an autologous or allogeneic stem cell transplant in the previous 365 days
* Requires a bronchoalveolar lavage for clinical indications
* Signed consent Exclusion criteria
* Lack of signed informed consent

Ages: 0 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients less than 30 years old who have had a hematopoietic stem cell transplantation and require a BAL for clinical diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2016-09-15 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage concordance between massively paralleled sequencing (MPS) and standard microbiological technique results. | 10 days
  Children, adolescents and young adult (CAYA) hematopoietic stem cell transplantation (HSCT) subjects with clinical symptoms/indications will undergo bronchoalveolar lavage (BAL), with samples from those with sufficient BAL fluid yield (>10ml) undergoing both massively paralleled sequencing and standard microbiological technique comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Rosenblum, MD, Principal Investigator — New York Medical College

IPD SHARING:
Plan to Share IPD: Yes
Will submit manuscript for peer-reviewed publication.
Supporting Information: CSR
Time Frame: submit for publication Q4 2019